CLINICAL TRIAL: NCT02497300
Title: Vascular Effects of Mineralocorticoid Receptor Antagonism in Kidney Disease
Acronym: VEMAKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Eric Judd, Assistant Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F140508008
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Chronic Kidney Disease; Albuminuria
Keywords: Mineralocorticoid Receptor Antagonists; Mineralocorticoid Effects
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria | interventions — Spironolactone; Amiloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spironolactone (Experimental): Participants will be randomized to spironolactone 25mg daily for the 1st or 2nd 6 week treatment period.
  Interventions: Drug: Spironolactone
- Amiloride (Active Comparator): Participants will be randomized to amiloride 5mg daily for the 1st or 2nd 6 week treatment period.
  Interventions: Drug: Amiloride

INTERVENTIONS:
Drug: Spironolactone
  Arms: Spironolactone
Drug: Amiloride
  Arms: Amiloride

SUMMARY:
Vascular endothelial dysfunction increases cardiovascular (CV) risk and contributes to the progression of chronic kidney disease (CKD). Mineralocorticoid receptor (MR) antagonists have been shown to improve endothelial function, as well as decrease CV mortality and proteinuria. The specific biochemical pathways that produce these pharmacological effects for MR antagonists, however, are poorly understood. This study investigates the effect of MR antagonism on endothelial function in patients with moderate (stage III) CKD using a randomized, controlled trial. Three specific aims are proposed: Aim 1: To determine if spironolactone improves endothelial function as compared to amiloride in patients with stage III CKD; Aim 2: To determine if oxidative stress is associated with changes in endothelial function by spironolactone compared to amiloride in patients with stage III CKD; and Aim 3: To determine if endothelial dysfunction contributes to albuminuria in patients with stage III CKD. The clinical relevance is to improve understanding of the mechanisms of kidney function decline in CKD in order to develop interventions to delay or prevent dialysis, which would translate into alleviating patient suffering, caregiver burden, and health care costs.

DETAILED DESCRIPTION:
Study participants with proteinuric, stage III CKD will be randomly assigned in a double-masked fashion to spironolactone 25mg daily or amiloride 5 mg daily for 6 weeks and then crossed over to the alternate study medication after a 1 month wash-out period. Vascular function will be assessed at baseline and the end of each 6 week treatment period by: 1) ultrasound guided flow-mediated dilation (FMD) of the brachial artery, 2) impedence cardiography, 3) pulse-wave velocity, 4) 24 hour ambulatory blood pressure monitoring, and 5) serum and urine biomarkers. Participants will undergo a total of 7 visits over 16-18 weeks; 3 of the 7 visits will involve vascular function testing.

A study visit where vascular function testing is to be performed will begin at 0800 in the morning and start with a vital sign assessment including height, weight, body fat percent, and left arm automated BP measurement followed by confirmation of fasting status and a brief past medical history. Each participant will then lie supine for 10 minutes in preparation for vascular function testing. Following the pulse wave velocity, impedence cardiography, and FMD measurements, the participant will have his/her blood and urine collected for laboratory testing. Laboratory testing will include ~20 mL of blood for plasma and serum testing. Participants will return 24 hour urine samples and have a 24 hour ambulatory monitor placed. This entire visit is expected to take 2 hours.

Study visits where vascular function testing will not be performed (e.g., screening visit, visit 2, visit 4, and visit 5; should last 30 minutes and involve a medication assessment, vital sign check, and blood collection for serum potassium (~4 mL of blood).

All study medication will be prepared by the the University of Alabama (UAB) Research Pharmacy in matching capsules and placed in pill bottles labeled "A" and "B". The order of medication dispensing will follow simple randomization using an a priori randomization list prepared by the research pharmacy. All study personnel with participant interaction are masked to the order of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years of age)
* CKD (eGFR 25-60 mL/min/1.73m2) with urine albumin-to-creatinine ratio > 30 mg/g
* CKD (eGFR > 60 mL/min/1.73m2) with urine albumin-to-creatinine ratio ≥ 300 mg/g

Exclusion Criteria:

* Severe hypertension (HTN) (office BP ≥ 160/100 mm Hg)
* Hypotension (office BP < 110/70 mm Hg)
* Serum potassium > 5 milliequivalent/L
* History of arrhythmia, including atrial fibrillation
* Pregnant or breast feeding woman
* Diabetes mellitus (DM) type 1
* Diabetes mellitus type 2 with glycosylated hemoglobin ≥ 6.5%
* Dementia or cognitive impairment prohibiting consent
* History of ischemic stroke, unstable angina, or myocardial infarction within the past 6 months
* Allergy or intolerance to spironolactone or amiloride
* Use of an MR antagonist or an epithelial sodium channel blocking medication within the last month
* Known primary aldosteronism or renal artery stenosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hypertension Research Clinic at UAB, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Spironolactone First, Then Amiloride: Participants will be randomized to spironolactone 25mg daily for the 1st treatment period of 6 weeks
  Spironolactone
- Amiloride First, Then Spironolactone: Participants will be randomized to amiloride 5mg daily for the 1st treatment period of 6 weeks
  Amiloride
Period: First Intervention (6 Weeks)
Arm/Group | Spironolactone First, Then Amiloride | Amiloride First, Then Spironolactone
Started | 13 | 6
Completed | 12 | 6
Not Completed | 1 | 0
Period: Washout (1 Month)
Arm/Group | Spironolactone First, Then Amiloride | Amiloride First, Then Spironolactone
Started | 12 | 6
Completed | 12 | 6
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Spironolactone First, Then Amiloride | Amiloride First, Then Spironolactone
Started | 12 | 6
Completed | 10 | 5
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Unable to meet recruitment goals
Groups:
- Spironolactone First, Then Amiloride: Randomized to 25mg daily of spironolactone as the first study medication.
- Amiloride First, Then Spironolactone: Randomized to 5mg daily of amiloride as the first study medication.
- Total: Total of all reporting groups
Arm/Group | Spironolactone First, Then Amiloride | Amiloride First, Then Spironolactone | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 6 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (15.7) | 47.5 (17.4) | 47.6 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 6 | 0 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Difference in 24 Hour Ambulatory Systolic Blood Pressure
Description: The study was not able to meet its recruitment goal, and participant numbers were too low to test the intended primary outcome of "Difference in percent change of ultrasound-guided flow-mediated dilation between 6 weeks of spironolactone vs. 6 weeks of amiloride." The change in 24hr ABPM systolic BP (Baseline - 6 week) is reported here.
Time Frame: 6 weeks
Population: Some participants had missing or incomplete 24 hour ambulatory blood pressure monitoring
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Spironolactone Exposure: After 6 weeks of spironolactone 25mg daily (combined first or second treatment period)
- Amiloride Exposure: After 6 weeks of amiloride 5mg daily (combined first or second treatment period)
Arm/Group | Spironolactone Exposure | Amiloride Exposure
Number analyzed (Participants) | 16 | 16
mm Hg | 7.7 (18.4) | 12.5 (23.3)

2. Primary Outcome: Change in Oxidative Stress as Measured by Urine Levels of F2-isoprostanes
Description: Difference in level of urine 8-iso-prostaglandin-F2-alpha per mg of creatinine levels between 6 weeks of spironolactone vs. 6 weeks of amiloride.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng F2 isoprostane/mg creatinine
Groups:
- Spironolactone: Randomized to 25mg daily of spironolactone as the first study medication.
- Amiloride: Randomized to amiloride 5mg daily as the first study medication
Arm/Group | Spironolactone | Amiloride
Number analyzed (Participants) | 10 | 5
ng F2 isoprostane/mg creatinine | -2.77 (6.3) | -0.17 (0.2)

3. Primary Outcome: Change in Albuminuria
Description: Change of the urine albumin-to-creatinine ratio (baseline - post-study med) after 6 weeks of spironolactone vs. 6 weeks of amiloride.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg albumin/g creatinine
Arm/Group | Spironolactone | Amiloride
Number analyzed (Participants) | 10 | 5
mg albumin/g creatinine | 129 (326) | 285 (565)

4. Secondary Outcome: Change in Serum Potassium
Description: Difference in serum potassium levels (baseline - post-medication) after 6 weeks of spironolactone vs. 6 weeks of amiloride.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Spironolactone | Amiloride
Number analyzed (Participants) | 10 | 5
mEq/L | 0.4 (1.5) | -0.5 (0.6)

5. Secondary Outcome: Change in Serum Creatinine (Baseline - Post-medication)
Description: Difference in serum creatinine (baseline - post-medication) after 6 weeks of spironolactone vs. 6 weeks of amiloride.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Spironolactone | Amiloride
Number analyzed (Participants) | 10 | 5
mg/dL | 0.2 (0.8) | -0.1 (0.3)

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Amiloride First, Then Spironolactone: Randomized to amiloride 5mg daily as the first study medication
- Spironolactone Second Intervention: Received 25mg spironolactone after 4 week washout
- Amiloride Second Intervention: Received 5mg amiloride after 4 week washout
Arm/Group | Spironolactone First, Then Amiloride | Amiloride First, Then Spironolactone | Spironolactone Second Intervention | Amiloride Second Intervention
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 1/6 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spironolactone First, Then Amiloride (N=13) | Amiloride First, Then Spironolactone (N=6) | Spironolactone Second Intervention (N=6) | Amiloride Second Intervention (N=12)
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Serum potassium level > 6.0 mEq/L

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02497300/Prot_000.pdf